CLINICAL TRIAL: NCT04775654
Title: The Effects of Blackcurrant Supplementation on Eye Health: a Randomized, Double Blind, Placebo Controlled Clinical Trial
Brief Title: The Effects of Blackcurrant Supplementation on Eye Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: Artemis International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-02-7800
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Eye Strain; Eye Fatigue
Keywords: black currant; blackcurrant; Ribes nigrum; digital eye fatigue; eye health; computer vision syndrome; dietary supplement
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the individuals providing informed consent are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): Participants consume 455mg of blackcurrant extract standardized to contain 50mg anthocyanins in a 2-capsule dose for 70 days.
  Interventions: Dietary Supplement: Blackcurrant
- Placebo (Placebo Comparator): Participants consume 2 capsules of microcrystalline cellulose for 70 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Blackcurrant — Two capsules containing 455mg of CurrantCraft 11% black currant extract.
  Arms: Supplement
Other: Placebo — Two capsules containing an inert material.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential for supplementation with black currant to support eye health among otherwise healthy adult women who spend 6+ hours per day using digital screens.

DETAILED DESCRIPTION:
Women who are informed about the study and provide informed consent will be randomized to one of two groups: supplement and placebo. Group assignment will be a 1:1 ratio to supplement (455mg of blackcurrant standardized to 50mg anthocyanins in 2 capsules/day) or placebo (2 capsules/day). Outcomes will be assessed at baseline and again on day 70.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 30-60
* Lives in the United States
* Employed full time in an online work environment OR enrolled full time in an online learning environment (average of 6+ hours per day)
* Ability to understand study instructions
* Ability to provide informed consent
* Residence within 100 miles of the study center

Exclusion Criteria:

* Low blood pressure
* Uncontrolled hypertension (i.e. systolic/diastolic blood pressure > 140/90)
* Uncontrolled diabetes (i.e. fasting blood glucose >180mg/dl)
* Any blood clotting disorder
* Ocular disease
* Best corrected visual acuity <20/30
* Cataracts
* Renal disease
* Active hepatitis or cirrhosis
* Acute or chronic infectious disease
* Pregnant
* Breastfeeding
* Currently trying to conceive
* Surgical or other invasive procedure planned within the intervention period

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 57 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ocular discomfort on day 70. | Baseline and day 70
  The Ocular Discomfort scale is a validated self reported instrument assessing ocular discomfort symptoms. The scale contains 6 domains with a combination of likert scale (ranging from 1-7) and dichotomous (yes/no) questions. Higher scores indicate greater visual fatigue.
Change from baseline in visual fatigue on day 70. | Baseline and day 70
  The Visual Fatigue scale is a validated self reported instrument assessing visual fatigue symptoms. It is a 6-question scale which asks about immediate symptoms (such as dry eyes). Participants rank their symptoms on a likert scale scored from 1-7, with higher scores indicating more severe symptoms.
Change from baseline in computer vision symptoms on day 70. | Baseline and day 70
  The Computer Vision Symptom scale is a validated self reported instrument assessing computer vision symptoms. The scale measures 17 symptom domains, with scores ranging from 1-4 to 1-7. On each domain, higher scores indicate greater severity.
Change from baseline in symptoms of computer vision syndrome on day 70. | Baseline and day 70
  The Computer Vision Syndrome Questionnaire is a validated self reported instrument assessing computer vision symptoms. The scale measures the presence or absence of 16 symptoms producing scores from 0-16. Higher scores indicate more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie R Hawkins, PhD, Principal Investigator — Franklin Health Research & Education Center
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No